CLINICAL TRIAL: NCT06688305
Title: 68Ga-NI-FAPI PET/CT: First-in-human Study in Patients With Various Cancers
Brief Title: 68Ga-NI-FAPI PET/CT: First-in-human Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-68Ga-NI-FAPI
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NI-FAPI PET/CT (Experimental): PET/CT imaging in patients with malignant tumors: each patient underwent a PET/CT scan after intravenous administration of 68Ga-NI-FAPI.
  Interventions: Drug: 68Ga-NI-FAPI

INTERVENTIONS:
Drug: 68Ga-NI-FAPI — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-NI-FAPI.

SUMMARY:
68Ga-NI-FAPI is a novel radiotracer incorporating a hypoxia sensitive nitroimidazole (NI)-moiety and a FAP-targeting. In this study, we observed the safety, biodistribution, radiation dosimetry and diagnostic value of 68Ga-NI-FAPI PET/CT in patients with different types of cancer.

DETAILED DESCRIPTION:
Carcinoma-associated fibroblasts (CAFs) are an integral part of the tumor microenvironment, and fibroblast activation protein (FAP), as a specific marker of CAFs, is overexpressed in more than 90% of epithelial malignant tumors' CAFs, with limited expression in normal tissues, making it an appropriate target for various tumors. Currently, several tracers targeting FAP for diagnostic purposes have been developed, such as 68Ga-FAPI-04, 68Ga-FAPI-02, and showed high efficacy in tumor staging and restaging. 68Ga-NI-FAPI is a novel agent incorporating a hypoxia sensitive nitroimidazole (NI)-moiety and a FAP-targeting. This pilot study was prospectively designed to evaluate the safety, biodistribution, radiation dosimetry and diagnostic value of 68Ga-NI-FAPI in patients with different types of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Various solid tumors with available histopathological findings
* Signed informed consent

Exclusion Criteria:

* pregnant or lactational women
* who suffered from severe hepatic and renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability | up to 1 week
  Hematologic status, liver function, renal function and General vital signs were recorded before and 1 week after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Dosimetry of normal organs and tumors | From right after tracer injection to 150 minutes at post-injection
  The semiquantitative dosimetry will be performed based on PET/CT acquisitions after the first administration of 68Ga-NI-FAPI. The dose delivered to normal organs and tumors will be recorded.

OTHER OUTCOMES:
Diagnostic value | through study completion, an average of 3 months
  Sensitivity and Specificity of 68Ga-NI-FAPI for patients with various cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Zang J, Cheng H, Luo Y, Jin W, Lai Y, Zheng Q, Peng Y, Kung HF, Zhu L, Ke C, Liu C, Miao W. First-in-human study of a novel bifunctional PET tracer [68Ga]Ga-DOTA-NI-FAPI-04 targeting FAP and hypoxia. Eur J Nucl Med Mol Imaging. 2025 Oct 31. doi: 10.1007/s00259-025-07625-0. Online ahead of print. PMID 41168395